CLINICAL TRIAL: NCT00016653
Title: A Multicenter Randomized Placebo-controlled Double-blind Study to Assess Efficacy and Safety of Glutamine and Creatine Monohydrate in Duchenne Muscular Dystrophy
Brief Title: Creatine and Glutamine in Steroid-Naive Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cooperative International Neuromuscular Research Group (Network)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CNMC0599
Record Dates: First submitted 2001-05-21; First posted 2001-05-23 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: Duchenne; muscular; dystrophy; treatment
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Creatine; Glutamine

INTERVENTIONS:
Drug: Creatine Monohydrate
Drug: Glutamine

SUMMARY:
This study will help to determine the effectiveness of glutamine and creatine as a possible therapy for DMD. Boys with DMD who are enrolled in this trial will be randomly chosen to receive creatine monohydrate or glutamine or an inactive placebo orally for six months. Once a month during the six-month treatment period, the study participants will have their muscle strength evaluated using manual and computerized testing methods. This study will be conducted at several CINRG Centers throughout the U.S., Belgium, Israel and Puerto Rico. This study is supported by the Muscular Dystrophy Association.

DETAILED DESCRIPTION:
PURPOSE OF THE STUDY The purpose of this study is to see if children with Duchenne muscular dystrophy (DMD) who are given glutamine (a nutritional supplement) or creatine monohydrate (a nutritional supplement) have changes in strength compared to children who are given no medicinal treatment. Children who are chosen to be in this research study will be diagnosed with DMD, be between the ages of 5 and 10 years old, and will not have participated in any other DMD clinical trials within the last year, and will not have been on medications that disqualify them from participation in this trial. All children in this clinical trial are entered at the discretion of the doctors in charge of the study. During the first and second visits, children who fulfill the criteria for participation in the clinical trial will be determined. We expect 50 subjects to participate at CINRG centers worldwide.

PROCEDURES

Children will be randomized (a procedure like flipping a coin) into one of three groups: treated with glutamine, treated with creatine monohydrate, or untreated (placebo: a sugar pill with no medication). Neither parents, children, nor the doctors treating the children will know the group each child has been assigned to. Because of the study design, there is a possibility that children will receive no treatment (placebo group) during the clinical trial. During the trial children must take one supplement mixed with water in the morning and supplements mixed with water each night.

Nine (9) clinic visits are required to complete this clinical trial. During visits to the clinic, each child will be evaluated by members of the research team to determine the child?s strength. Strength will be measured in different ways: manual testing, quantitative testing, and the usual measures used during visits to the neurologist (child will be asked to rise from the floor, walk across room, etc.). Manual testing is the way strength is usually measured by your child?s doctor. The quantitative muscle strength test (QMT) is a mechanical way to measure strength: the child sits/lays on an examining table and is asked to pull/push a strap. This test will determine the strength of different muscle groups in kilograms of force. An electrocardiogram (ECG, a heart test) will be performed during screening visit 2 and month 6 and blood (a small amount equal to about 2 to 3 tablespoons) will be drawn on screening visit 2 and months 1, 3 and 6. Urine tests will be done at screening visit 2 nd months 1, 3 and 6 to monitor kidney function.

ELIGIBILITY:
INCLUSION CRITERIA

* Aged 5 - 9 years old
* Able to walk without assistance
* Diagnosis of DMD confirmed by one of the following:
* a) Positive X-linked family history; or
* b) Dystrophin immunofluorescence and/or immunoblot, which shows complete dystrophin deficiency, and clinical picture consistent with DMD; or
* c) Gene deletion test positive in the central rod domain (exons 25 - 60) of dystrophin, where reading frame can be predicted as 'out-of-frame', and clinical picture consistent with DMD.
* Glucocorticosteroid-naive (i.e. has not been treated with prednisone or deflazacort within 1 year before the study began), or has been involved in other therapeutic research protocol within the last year
* Forced Vital Capacity (a lung function test) > 50% of predicted value
* Evidence of muscle weakness by MRC score or clinical functional evaluation
* MRC (manual muscle test) score variability no greater than 10% between screening visits 1 and 2

EXCLUSION CRITERIA

* Failure to achieve any of the criteria listed above
* Symptomatic DMD carrier
* Symptomatic cardiomyopathy or ventricular arrhythmias
* Previous (6 months or less) or current use of glutamine or creatine (for DMD or any other indication)
* Use of carnitine, other amino acids, coenzyme Q10, or any herbal medicines within the last month
* History of significant concomitant illness or significant impairment of renal or hepatic function
* Evidence of allergy to chocolate or milk solids (substances will be delivered in a powdered hot cocoa mixture)

Ages: 5 Years to 9 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48
Dates: Start 2000-06; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Diana M Escolar, MD, Study Director — Cooperative International Neuromuscular Research Group; Gunnar Buyse, MD, PhD, Study Director — Cooperative International Neuromuscular Research Group
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Escolar DM, Buyse G, Henricson E, Leshner R, Florence J, Mayhew J, Tesi-Rocha C, Gorni K, Pasquali L, Patel KM, McCarter R, Huang J, Mayhew T, Bertorini T, Carlo J, Connolly AM, Clemens PR, Goemans N, Iannaccone ST, Igarashi M, Nevo Y, Pestronk A, Subramony SH, Vedanarayanan VV, Wessel H; CINRG Group. CINRG randomized controlled trial of creatine and glutamine in Duchenne muscular dystrophy. Ann Neurol. 2005 Jul;58(1):151-5. doi: 10.1002/ana.20523. PMID 15984021